CLINICAL TRIAL: NCT06237582
Title: Inferior Epigastric Lymp Node (IELN) Basin as a Possible Systemic Metastatic Pathway of Ovarian Peritoneal Metastases
Acronym: OvEpiLyPath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OvEpiLyPath
Record Dates: First submitted 2023-12-01; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-11

CONDITIONS: Carcinomatosis, Peritoneal
Keywords: epigastric lymph node; cytoreductive surgery; ovarian cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): patients planned for complete cytoreductive surgery
  Only one arm in the study: all patients operated for complete cytoreductive surgery and who signed informed consent form
  Interventions: Procedure: epigastric lymph node biopsy

INTERVENTIONS:
Procedure: epigastric lymph node biopsy — epigastric lymph node biopsy and analysis to evaluate rate dissemination of ovarian carcinomatosis by this way

SUMMARY:
The IELN basin could represent a primary LN relay for systemic metastatic dissemination in patients with OPM. This newly described lymphatic pathway of metastatic dissemination of OPM may be involved in certain presentations of peritoneal dissemination. The presence of invaded IELN may represent a new biomarker predictive of the pattern of progression of OPM and a related risk for systemic dissemination.

DETAILED DESCRIPTION:
Background:

More than two thirds of all patients with epithelial ovarian carcinoma have an advanced stage III or IV at diagnosis. However, in select group of patients, particularly in those with low tumor volume, parietal and visceral peritonectomy with the aim of complete macroscopic cytoreduction and hyperthermic intraperitoneal chemotherapy (HIPEC) is feasible and associated with a reasonable morbidity rate and mortality rate in patients with peritoneal carcinomatosis and ovarian cancer. The role of Peritoneal Cancer Index, expressing the tumor volume, was also found to be a prognostic indicator for the survival in these patients. A therapeutic approach that combined CRS + HIPEC could achieve long-term survival in selected groups of patients with ovarian peritoneal metastases (OPM) tumors with acceptable morbidity and mortality. A good expertise and a high volume of patients are necessary to manage PC and to further improve results.

Very few studies have explored the pathophysiological mechanisms of PM development and progression. The main mechanism of reported peritoneal dissemination that has been reported is a stepwise dissemination including the exfoliation of tumoral cells from the primary tumour into the peritoneal cavity. The pathophysiological mechanisms underlying systemic dissemination in patients presenting with PM are also poorly understood. The most well-known lymphatic dissemination pathways from the peritoneum into supra-diaphragmatic lymph nodes (LNs) are the retroperitoneal lymphatic pathway and the cardio-phrenic LNs. The presence of involved cardio-phrenic LNs is predictive of PM involvement. However, detection of these LNs is based on imaging that has a limited sensitivity (65%) and surgical access requires the opening of the diaphragm.

Recently, the investigators reported, for the first time, a new lymphatic route of systemic dissemination of PM. They reported LN metastases in the inferior epigastric LN basin (IELN). In this series, metabolic and morphologic imaging were not able to preoperatively predict the status of IELN. These LNs represent potential predictive factors of survival in patients treated for PM. The advantage of this LN basin is its easy surgical access that allows resection without increasing postoperative complications. The exact conditions for dissemination in IELN and their prognostic role remain undetermined.

The primary objective of this study is to evaluate the incidence of IELN basin involvement in patients with PM undergoing complete CRS. The secondary objectives are to evaluate the capacity of preoperative imaging to detect these lesions and to define conditions for IELN involvement.

Hypotheses of the research:

The IELN basin could represent a primary LN relay for systemic metastatic dissemination in patients with OPM. This newly described lymphatic pathway of metastatic dissemination of OPM may be involved in certain presentations of peritoneal dissemination. The presence of invaded IELN may represent a new biomarker predictive of the pattern of progression of OPM and a related risk for systemic dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo complete cytoreductive surgery for peritoneal metastases from ovarian origin

Exclusion Criteria:

* Minor patients
* Patients unable to give written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the incidence of IELN invasion by ovarian cancer | 2 years
  Histopathological analysis of concerned lymph nodes, with or without immunohistochemical profiling when needed.
  Identification of metastatic disease (ovarian cancer), present in the inferior epigastric lymph nodes basin

SECONDARY OUTCOMES:
Evaluation of the proportion of invaded IELN | 2 years
  Assess the incidence (in %) of IELN involvement with metastatic ovarian cancer, with respect to the patient's PCI and the peritoneal zones involved mostly by the disease (Sugarbaker zones), e.g. pelvic peritoneum versus flanks, versus upper abdominal quadrants.
In cases of IELN positivity, review thoroughly preoperative scans and MRIs in order to detect radiological features, usually overlooked, that could help identify the positivity of these LNs prior to pathological analysis. | 2 years
  comparison of imaged IELN and pathological analysis

CONTACTS AND LOCATIONS:
Overall Officials: Antoine El Asmar, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium